CLINICAL TRIAL: NCT05815329
Title: Validation and Clinical Usability of a New Screening Tool: MASCoD - Multidimensional Assessment of Subjective Cognitive Decline
Brief Title: MASCoD - Multidimensional Assessment of Subjective Cognitive Decline
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2666
Record Dates: First submitted 2023-03-13; First posted 2023-04-18 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Cognitive Decline
Keywords: mild cognitive impairment; subjective cognitive decline; neuropsychological rehabilitation
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: randomised controlled clinical study with follow up (experimental group and waiting list)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rehabilitation group (Experimental): Outpatients undergoing neurorehabilitation through Neurotablet
  Interventions: Other: cognitive training
- waiting list (No Intervention): Outpatients not undergoing rehabilitation during the study. They will have the possibility to carry on the rehabilitation at the end of the study

INTERVENTIONS:
Other: cognitive training — After the multidimensional evaluation at T0, the participants will be randomly allocated into an experimental group and a wait list control group. Specifically, cognitive training will be offered to half of the outpatients included in this research by means of technological devices (Neurotablet). A neuropsychologist will supervise the cognitive training offline (about 30 minutes per 5 days, 8 weeks) and through a face-to-face 1 hour-session each week per each outpatient.
  Arms: rehabilitation group

SUMMARY:
Subjective cognitive decline-SCD is a subclinical cognitive impairment subjectively experienced without being detectable from a diagnostic and neuropsychological perspective. It can negatively impact on patient's frailty and quality of life and it may be prodromal to severe cognitive impairment. Currently, only a few screening tools focusing mainly on memory complaints exist.

The aim of this study is to analyze if a new screening tool called MASCoD (Multidimensional Assessment of Subjective Cognitive Decline) can detect and monitor the SCD, predicting the risk of developing severe cognitive decline over time.

Specifically, the investigators have the following aims:

primary objectives:

1. To assess the construct validity and tune the clinical cutoffs of the new instrument through the correlation of MASCoD scores with neuropsychological evaluation and brain 18F-FDG-PET.
2. To assess the clinical validity (predictive capability) of the new instrument through a classification model (dependent variable: brain 18F-FDG-PET examination; independent variable: MASCoD; control variables: gender, age and neuropsychological evaluation).

Secondary objective:

To evaluate the suitability of MASCoD as tool for the monitoring of patients over time. Specifically, the investigators want to evaluate if the MASCoD score is able to assess the effects of a cognitive treatment and, in turn, to identify outpatients who most likely will benefit from it.

After the multidimensional evaluation at T0, the participants will be randomly allocated into an experimental group and a wait list control group. Specifically, cognitive training will be offered by means of technological devices (Neurotablet).

At T1, all outpatients (experimental group and wait list control group) will be evaluated through MASCoD and the extensive neuropsychological evaluation for the second time.

DETAILED DESCRIPTION:
Subjective cognitive decline (SCD) is a subclinical cognitive impairment, which is complained by the individual without being objectively supported at diagnostic and neuropsychological levels. It can negatively influence outpatient's frailty and quality of life, as well as caregiver's burden. It may be associated with anxious and/or depressive symptoms too. Moreover, it can be prodromal to Mild Cognitive Impairment or dementia. Concerning this issue, to date, imaging biomarkers (e.g. positron emission tomography - brain 18F-FDG-PET), can be considered a promising method to predict the development of different forms of future cognitive decline. However, this examination is very expensive for the healthcare system.

Although the clinical manifestations of SCD can differ along several cognitive domains (e.g. memory problems, mental slowness and concentration difficulties, self-perceived deterioration in usual cognitive performance), as far as the investigators know, there are currently only screening tools to investigate subjective memory complaints.

Rehabilitation can play a pivotal role in this condition and non-pharmacological interventions on SCD, as cognitive training, could maintain on existing cognitive resources and slow the rate of possible increasing cognitive decline. To date, lower-functioning individuals seem to benefit more from cognitive training, in particular concerning working memory and executive functions (i.e. inhibition).

Thus, a screening tool assessing all possible subclinical manifestations of SCD and risk factors is needed to support professionals in making differential diagnosis and to predict the risk of developing severe cognitive impairment over time, proposing a personalized care path. From a clinical and research standpoint, a useful screening tool is expected to be brief for usual clinical assessment and research protocol, as well as administrable by different professionals and in various healthcare settings. Moreover, it should suggest targeted interventions to maximize the psychophysical outcome. The development of such a screening tool would address the current shortage of rapid, economic and validated instruments globally assessing over time cognition affected by this condition.

In light of the above issues, the investigators propose a brief, not expensive, multidimensional screening tool called MASCoD (Multidimensional Assessment of Subjective Cognitive Decline) developed on the basis of literature and the clinical experience provided by an experts' panelist (i.e. psychologists, neuropsychologists, neurologists) employed at the Institute for Research, Hospitalization and Healthcare (IRCCS) - Istituti Clinici Scientifici (ICS) Maugeri - Institute of Montescano and Pavia, Italy. It is composed of a general form for socio-demographic data and the following sections: a) risk factors for SCD; b) memory and executive symptoms; c) anxious/depressive or distressing symptoms. There are four increasing risk levels (i.e. low, medium with emotional complaints, medium without emotional complaints, high risk) of developing a severe cognitive impairment. Two versions of MASCoD have been proposed: one for the first baseline screening and one for the follow up assessments.

The aim of this study is to analyze if MASCoD can detect and monitor the SCD, predicting the risk of developing severe cognitive decline over time.

Specifically, the investigators have the following aims:

primary objectives:

1. To assess the construct validity and tune the clinical cutoffs of the new instrument through the correlation of MASCoD scores with neuropsychological evaluation and brain 18F-FDG-PET.
2. To assess the clinical validity (predictive capability) of the new instrument through a classification model (dependent variable: brain 18F-FDG-PET examination; independent variable: MASCoD; control variables: gender, age and neuropsychological evaluation).

Secondary objective:

To evaluate the suitability of MASCoD as tool for the monitoring of patients over time. Specifically, the investigators want to evaluate if the MASCoD score is able to assess the effects of a cognitive treatment and, in turn, to identify outpatients who most likely will benefit from it.

Eligible patients will be selected among consecutive outpatients requiring a neurological assessment for possible SCD at: a) ICS) Maugeri - Institute of Montescano, Neurophysiopatology Unit (DTCP - Diagnostic-Therapeutic Care Pathway for dementia), b) Neurology Unit Neurology Unit, Civil General Hospital in Voghera (PV) ASST Pavia, c) Rehabilitation Department Voghera Stradella Mortara (PV) Hospital ASST di Pavia.

The inclusion criteria are the following: reported SCD without any other cognitive or neurological issue, Italian education, adult (> 55 years old), understanding of research aims, signed informed consent, participation on a voluntary and non-retributed bases.

The exclusion criteria are the following: serious clinical conditions (e.g. severe cardiac and respiratory problems, neoplasia) and prior diagnosis of psychiatric disorders according to DSM-5, prior diagnosis of cognitive decline, relevant visuo-perceptive or hearing deficits, illiteracy or relapse in illiteracy, refusal to partake into the research.

Form a methodological point of view, outpatients will undergo an extensive neuropsychological evaluation, brain 18F-FDG-PET, as required by the Maugeri DTCP for cognitive disorders.

After the multidimensional evaluation at T0, the participants will be randomly allocated into an experimental group and a wait list control group. Specifically, cognitive training will be offered to half of the outpatients included in this research, by means of technological devices (Neurotablet). A neuropsychologist will supervise the cognitive training offline (about 30 minutes per 5 days) and through a face-to-face 1 hour-session each week per each outpatient. The wait list control group will only perform neuropsychological assessment at the 6-month follow-up, without any treatment between T0 and T2. The latter will then be able to perform the same cognitive stimulation training subsequent to the control group and follow-up evaluation.

At T1, all outpatients (experimental group and wait list control group) will be evaluated through MASCoD and the extensive neuropsychological evaluation for the second time (6 months- 1 year).

ELIGIBILITY:
Inclusion Criteria:

* reported subjective cognitive decline without any other cognitive or neurological issue,
* Italian education,
* adult (> 55 years old),
* understanding of research aims,
* signed informed consent,
* participation on a voluntary and non-payied bases.

Exclusion Criteria:

* serious clinical conditions (e.g. severe cardiac and respiratory problems, neoplasia)
* prior diagnosis of psychiatric disorders according to DSM-5,
* prior diagnosis of cognitive decline,
* relevant visuo-perceptive or hearing deficits,
* illiteracy or relapse in illiteracy,
* refusal to partake in the research.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-08-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
instrument validation | baseline
  To assess the construct and clinical validity, and tune the clinical cutoffs of the new instrument MASCoD

SECONDARY OUTCOMES:
screening for rehabilitation suitability | immediately after the cognitive training
  To evaluate the suitability of MASCoD as tool for the monitoring of patients over time. Specifically, the investigators want to evaluate if the MASCoD score is able to assess the effects of a cognitive treatment and, in turn, to identify outpatients who most likely will benefit from it.

CONTACTS AND LOCATIONS:
Locations (1):
- ICS Maugeri Montescano Institute, Montescano, Pavia, Italy